CLINICAL TRIAL: NCT05409625
Title: 3D Scanning and Transillumination vs Conventional Examination to Assess Caries Progression, Stability or Regression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Protocol MKR
Record Dates: First submitted 2021-12-16; First posted 2022-06-08 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Dental Caries
Keywords: 3D Scanner; Fluorescence; Transillumination; Dental Caries; Intraoral Scanner
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Young adults (Experimental): Participants aged between 18 and 30 years old without chronic diseases but with two caries lesions or more
  Interventions: Device: Intraoral Scanner (TRIOS 4, 3Shape TRIOS A/S, Copenhagen, Denmark); Device: Intraoral camera (DIAGNOcam, KaVo, Biberach, Germany, software version 3.0.1/2.9.1); Device: X-ray device (X-ray device SOREDEX, MINRAY®; Image plates VistaScan; Image plate scanner VistaScan Mini View, Dürr Dental); Procedure: Oral cleaning

INTERVENTIONS:
Device: Intraoral Scanner (TRIOS 4, 3Shape TRIOS A/S, Copenhagen, Denmark) — Intraoral scanner which is able to generate a 3D-model of the teeth and is being used for caries detection.
Device: Intraoral camera (DIAGNOcam, KaVo, Biberach, Germany, software version 3.0.1/2.9.1) — Intraoral camera used for caries detection in the occlusal and proximal surfaces.
Device: X-ray device (X-ray device SOREDEX, MINRAY®; Image plates VistaScan; Image plate scanner VistaScan Mini View, Dürr Dental) — X-ray device used for caries detection. Two radiographs (bitewings) are taken, one in each side.
Procedure: Oral cleaning — Removal of tartar and plaque. Tartar removal done at baseline and the fifth visit, but only on selected teeth at the second, third and fourth visit. Regular cleaning with a toothbrush done at all visits.

SUMMARY:
The objective of this study is to investigate whether the 3D scanner and accompanying software, as well as the transillumination method, can identify changes in primary caries lesions in caries-active patients, where selected lesions achieve a higher degree of plaque control than others over an 8-month period.

The working hypothesis of this study is that the two methods, scanning and transillumination, are as good as the traditional method (clinical examination complemented by radiographs) to assess whether caries lesions are progressing, stable or regressing. Progression, stability or regression of selected caries lesions are thus the endpoint, and the rationale is to investigate whether more objective measures can replace/supplement a subjective method to assess progression, stability or regression of caries lesions.

DETAILED DESCRIPTION:
Caries is a non-infectious disease of the hard tissues of the teeth that occurs with very high prevalence around the world. The aetiology and pathogenesis of the disease are well understood. Bacterial accumulation on the teeth (dental plaque) concomitant with the ingestion of fermentable carbohydrates promotes acid production deep within the plaque, which progressively demineralizes the underlying hard dental tissue. Caries thus involves mineral loss from the first crystal disintegrating (not clinically identifiable) through gradually increased demineralization, with the mineral loss being identified early by the tooth tissue changing colour, through the physical appearance of a fracture (cavity) in the tooth, to the complete damage of the tooth. Demineralization can be halted or controlled by daily brushing with fluoride toothpaste, provided that brushing, possibly supplemented with flossing, is carried out as demonstrated by dentists or dental hygienists. Adding professional cleaning, i.e. plaque removal with rotary brushes and flossing and performed by dentists/ dental hygienists or clinic assistants, e.g. once a month, can ensure that the lesion is stopped if daily home dental care is not optimal. If caries has occurred, it can be treated non-operatively or surgically, complemented by risk-related initiatives.

Caries can develop in relation to previously placed fillings. This is referred to as secondary caries. In contrast, the term primary caries is used for caries located on unfilled/restored areas of the tooth or its root surfaces. Whether primary or secondary, caries lesions' severity is classified as superficial, moderate or extensive. The last two diagnoses usually require operative treatment, i.e. a filling, or root canal treatment or extraction.

Caries is detected and diagnosed using a number of methods, the most common being a clinical visual/tactile examination of the teeth, complemented by radiographs. However, this method is highly subjective, and thus with large variation among dentists and dental hygienists, resulting in different treatment strategie. In addition, radiographs lack sensitivity in terms of detection of the initial caries lesions.

Researchers have therefore developed various devices and methods for a more objective modulation of mineral loss, including monitoring of individual caries lesions. Perhaps best known is the QLF (Quantitative Light Fluorescence) system, which uses fluorescence measurements of the tooth's response to demineralization. The latest technology using fluorescence for caries detection and classification is the intraoral 3D scanner with the integrated automated caries registration system, which has been developed and now for a few years has been tested in both in vitro and in vivo studies at the Department of Odontology of the University of Copenhagen (OI).

The technique is based on the fact that healthy and demineralized tooth tissue absorbs the blue-violet light (wavelength ~415 nm) and emits back fluorescent light with different light intensities, from bright green to brownish to red. In terms of detection and classification of caries lesions on occlusal surfaces, the scanner has overall a better reproducibility and a comparable accuracy expressed through sensitivity and specificity compared to a combination of the clinical and radiological examination.

Another method that has been widely investigated for the detection of initial proximal (between teeth) and occlusal caries lesions, without the use of ionizing radiation, is transillumination with near-infrared light (wavelength ~780 nm). In the transillumination method, the light is transmitted through the dental tissue. The caries lesions appear dark, like shadows, due to the scattering and absorption of the light in the porous demineralized tissue. In contrast, the healthy, transparent enamel tissue appears brighter as light penetrates this tissue with very low light scatter and almost no light absorption. This method is used by the intraoral camera "DIAGNOcam" (KaVo, Biberach, Germany) and has also been investigated by researchers from the Department of Odontology at the University of Copenhagen and 3Shape (3Shape TRIOS A/S, Copenhagen, Denmark) for implementation in the 3D intraoral scanner system. This has shown improved sensitivity in detecting initial approximal caries lesions that can be treated with preventive, non-operative methods.

One of the areas that remain to be investigated regarding the usefulness of the 3D scanner and transillumination camera as a caries diagnostic method is the monitoring of caries lesions between two or more examinations in the clinic, including how the systems respond to lesions that have received intensive treatment to stop their progression.

Method:

18-30-year-old young adults in Denmark with high caries activity. Potential participants are found by advertising for caries-active patients in the daily press, on the OI website or an announcement board at the OI.

When contacting a potential participant, information is provided about the study, in addition to what is stated in the advertisement, on the website or on announcement boards. After that the a clinical screening is conducted.

Participants (n ~33) are offered common caries prevention initiatives: improved self-care, toothbrush instruction using 1450 ppm fluoride toothpaste, dietary advice and topical fluoride treatment. In addition, selected superficial caries lesions on individual participants will be professionally cleaned once a month.

Study participants will receive dental check-ups at shorter intervals (approximately every 1.5 months) compared to standard treatment.

Participants with lesions requiring restorative treatment (media/profound lesions) or with teeth that must be extracted due to caries will be treated at the OI according to the usual rules.

A traditional clinical and radiological examination also includes the diagnosis of other pathological conditions of the oral cavity, which, if identified, will be treated at the OI, according to the usual rules, or the participant will be referred to a private dentist. Other diseases of the teeth and supporting tissues likely to be diagnosed in 18- to 30-year-olds are gingivitis, erosions and wisdom teeth which only partially emerge into the oral cavity (dentis retentus).

The examination shall be carried out at the Department of Odontology, University of Copenhagen (OI) First visit (Baseline) i) Relevant medical history. ii) Records: tooth and filling status (chart), as well as clinical plaque and gingival index ad modem Løe & Silness (1963) on selected teeth: 6+, 3+, 1+, +2, +4, +7, 7-,5-, 2-, -1, -3, -6.

iii) X-rays: 2 BW (X-ray device SOREDEX, MINRAY®; Image plates VistaScan; Image plate scanner VistaScan Mini View, Dürr Dental) with special holders for reproducible images.

iv) Dental cleaning and professional plaque removal, including flossing. v) 3D scanning vi) Transillumination method vii) ICDAS (International Caries Detection and Assessment System) registration viii) Treatment plan. ix) Treatment. Second visit (1.5 months) 3D intraoral scanning and ICDAS registration. Third visit (3 months) As at baseline, but no radiographs (BW). Fourth visit (~6 months) 3D intraoral scan and ICDAS registration. Fifth visit (8 months) As at 1st visit

In addition, participants will need to come a number of times to have their caries lesions that require restorative treatment treated.

At each visit, also when lesions are treated with fillings, polishing of selected lesions will be performed.

Monitoring plan The monitoring plan will be carried out in accordance with the standard procedures for clinical research at the Department of Odontology, University of Copenhagen.

Dental student Maria K. Riis will be responsible for daily data handling, secure data archiving, and recruitment of study participants.

Staff will be responsible for the overall monitoring of the study. This person (monitor) will soon be appointed by the Department of Odontology and will be responsible for a monthly check of the progress of the study, including the following parameters:

1. Verification of the presence of the consent form.
2. Verification that participants meet inclusion and exclusion criteria.
3. Verification of data collected versus source data.
4. Compliance with the protocol and documentation of any deviations

The reason for selecting participants aged 18 to 30 years is that they are more likely to have primary caries lesions (which is the focus area) than secondary caries lesions. In addition, other dental and oral diseases requiring treatment, such as extensive tooth wear, are less likely to be found during the traditional clinical and radiological examination conducted for the study in 18- to 30-year-olds compared to older individuals.

In addition, patients with chronic medical diseases or impaired salivary secretion are excluded as they are expected to have more extensive dental problems, which are not the focus of this study.

Publication of results The study protocol will be registered at www.ClinicalTrials.gov. The study results will be published in international scientific journals under the terms of the research agreement (09.01 Research collaboration agreement CPH (Copenhagen) University), to which this document is Appendix 2. This applies to negative, positive or inconclusive results. If contrary to expectations, publication in national/international journals is unsuccessful, the investigators will ensure, under the terms of the research agreement (09.01 Research collaboration agreement CPH University), that the data are published on the department's website. The research agreement (09.01 Research collaboration agreement CPH University) states that 3Shape can request that manuscript submission be postponed by up to three (3) months from the date of receipt, provided 3Shape proves that the postponement is important for 3Shape's prospects of acquiring intellectual property rights protection of the knowledge that the University has. The disclosure of knowledge shall always be made in compliance with the obligation of professional secrecy. The research agreement (09.01 Research collaboration agreement CPH University) states that 3Shape will use the anonymized clinical data for product development, regulatory and commercial activities related to 3Shape's products.

ELIGIBILITY:
Inclusion Criteria:

* Medically healthy young adult patients (18-30 years old) where individuals must have ≥ 20 teeth.
* Two or more active caries lesions

Exclusion Criteria:

* Patients with impaired salivary secretion
* Patients with chronic medical diseases.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2022-09-19 (Actual)

PRIMARY OUTCOMES:
1st Scanner caries score | Baseline
  Caries score registered using the intraoral scanner and the accompanying software (Trios, 3Shape TRIOS A/S, Denmark) which will provide an automated caries score. Scale used: 0 (sound surfaces), 1. (initial caries lesions in enamel or into the outer third of dentin), 2. (moderate - extensive caries lesions located into the middle - inner third of dentin).
2nd Scanner caries score | 1.5 months after baseline
  Caries score registered using the intraoral scanner and the accompanying software (Trios, 3Shape TRIOS A/S, Denmark) which will provide an automated caries score. Scale used: 0 (sound surfaces), 1. (initial caries lesions in enamel or into the outer third of dentin), 2. (moderate - extensive caries lesions located into the middle - inner third of dentin).
3rd Scanner caries score | 3 months after baseline
  Caries score registered using the intraoral scanner and the accompanying software (Trios, 3Shape TRIOS A/S, Denmark) which will provide an automated caries score. Scale used: 0 (sound surfaces), 1. (initial caries lesions in enamel or into the outer third of dentin), 2. (moderate - extensive caries lesions located into the middle - inner third of dentin).
4th Scanner caries score | 6 months after baseline
  Caries score registered using the intraoral scanner and the accompanying software (Trios, 3Shape TRIOS A/S, Denmark) which will provide an automated caries score. Scale used: 0 (sound surfaces), 1. (initial caries lesions in enamel or into the outer third of dentin), 2. (moderate - extensive caries lesions located into the middle - inner third of dentin).
5th Scanner caries score | 8 months after baseline
  Caries score registered using the intraoral scanner and the accompanying software (Trios, 3Shape TRIOS A/S, Denmark) which will provide an automated caries score. Scale used: 0 (sound surfaces), 1. (initial caries lesions in enamel or into the outer third of dentin), 2. (moderate - extensive caries lesions located into the middle - inner third of dentin).
1st NIR (Near-Infrared) caries score | Baseline
  Near-Infrared transillumination images of the premolar and molar teeth will be taken in order to examine the proximal and occlusal surfaces for possible caries lesions.
  (Score as 0-4: 0 (No caries. No dark gray area visible on approximal surface), 1 (Caries limited to enamel without any contact to the DEJ), 2 (Enamel caries with single-point contact to the DEJ), 3 (Enamel caries with extensive contact to the DEJ), 4 (Caries visible in enamel and dentin).
2nd NIR (Near-Infrared) caries score | 8 months after baseline
  Near-Infrared transillumination images of the premolar and molar teeth will be taken in order to examine the proximal and occlusal surfaces for possible caries lesions.
  (Score as 0-4: 0 (No caries. No dark gray area visible on approximal surface), 1 (Caries limited to enamel without any contact to the DEJ), 2 (Enamel caries with single-point contact to the DEJ), 3 (Enamel caries with extensive contact to the DEJ), 4 (Caries visible in enamel and dentin).
1st X-ray caries score | Baseline
  ICDAS grades caries radiologically as no radiolucency visible=0; radiolucency in outer 1/2 of enamel=1; radiolucency in inner 1/2 of enamel ±enamel dentin border=2; radiolucency in outer 1/3 of dentin=3; radiolucency in middle 1/3 of dentin=4; and radiolucency in inner 1/3 of dentin=5.
2nd X-ray caries score | 8 months after baseline
  ICDAS grades caries radiologically as no radiolucency visible=0; radiolucency in outer 1/2 of enamel=1; radiolucency in inner 1/2 of enamel ±enamel dentin border=2; radiolucency in outer 1/3 of dentin=3; radiolucency in middle 1/3 of dentin=4; and radiolucency in inner 1/3 of dentin=5.
1st Clinical ICDAS score | Baseline
  ICDAS registration graded as 0 = sound, brownish lesion < 1 mm = 1b, brownish lesion ≥ 1mm = 2b, whitish lesion after drying = 1w, whitish lesion without drying = 2w, fracture limited to enamel = 3, shadowing = 4, fracture exposing dentin but fracture less than ½ of extent of surface = 5, 6 as 5 but fracture ≥ ½ of extent of surface.
2nd Clinical ICDAS score | 1.5 months after baseline
  ICDAS registration graded as 0 = sound, brownish lesion < 1 mm = 1b, brownish lesion ≥ 1mm = 2b, whitish lesion after drying = 1w, whitish lesion without drying = 2w, fracture limited to enamel = 3, shadowing = 4, fracture exposing dentin but fracture less than ½ of extent of surface = 5, 6 as 5 but fracture ≥ ½ of extent of surface.
3rd Clinical ICDAS score | 3 months after baseline
  ICDAS registration graded as 0 = sound, brownish lesion < 1 mm = 1b, brownish lesion ≥ 1mm = 2b, whitish lesion after drying = 1w, whitish lesion without drying = 2w, fracture limited to enamel = 3, shadowing = 4, fracture exposing dentin but fracture less than ½ of extent of surface = 5, 6 as 5 but fracture ≥ ½ of extent of surface.
4th Clinical ICDAS score | 6 months after baseline
  ICDAS registration graded as 0 = sound, brownish lesion < 1 mm = 1b, brownish lesion ≥ 1mm = 2b, whitish lesion after drying = 1w, whitish lesion without drying = 2w, fracture limited to enamel = 3, shadowing = 4, fracture exposing dentin but fracture less than ½ of extent of surface = 5, 6 as 5 but fracture ≥ ½ of extent of surface.
5th Clinical ICDAS score | 8 months after baseline
  ICDAS registration graded as 0 = sound, brownish lesion < 1 mm = 1b, brownish lesion ≥ 1mm = 2b, whitish lesion after drying = 1w, whitish lesion without drying = 2w, fracture limited to enamel = 3, shadowing = 4, fracture exposing dentin but fracture less than ½ of extent of surface = 5, 6 as 5 but fracture ≥ ½ of extent of surface.
1st Caries activity assessment score | Baseline
  The activity of the clinically identified caries lesions (active/arrested) will be based on:
  Localisation of the lesion (No plaque stagnation area = 0, Plaque stagnation area = 1); Colour of the lesion (Brownish = 0; Whitish = 1); Feeling with probe (Lesion Smooth = 0; Lesion Rough = 1); No breakdown/breakdown on enamel surface: (No breakdown, or breakdown with smooth border area = 0; Breakdown with rough border area = 1); In case of gingival or proximal lesions (Healthy gingiva = 0; Bleeding on probing = 1).
  Arrested lesions total score ≤ 2 points; Active lesions total score > 2 points.
2nd Caries activity assessment score | 1.5 months after baseline
  The activity of the clinically identified caries lesions (active/arrested) will be based on:
  Localisation of the lesion (No plaque stagnation area = 0, Plaque stagnation area = 1); Colour of the lesion (Brownish = 0; Whitish = 1); Feeling with probe (Lesion Smooth = 0; Lesion Rough = 1); No breakdown/breakdown on enamel surface: (No breakdown, or breakdown with smooth border area = 0; Breakdown with rough border area = 1); In case of gingival or proximal lesions (Healthy gingiva = 0; Bleeding on probing = 1).
  Arrested lesions total score ≤ 2 points; Active lesions total score > 2 points.
3rd Caries activity assessment score | 3 months after baseline
  The activity of the clinically identified caries lesions (active/arrested) will be based on:
  Localisation of the lesion (No plaque stagnation area = 0, Plaque stagnation area = 1); Colour of the lesion (Brownish = 0; Whitish = 1); Feeling with probe (Lesion Smooth = 0; Lesion Rough = 1); No breakdown/breakdown on enamel surface: (No breakdown, or breakdown with smooth border area = 0; Breakdown with rough border area = 1); In case of gingival or proximal lesions (Healthy gingiva = 0; Bleeding on probing = 1).
  Arrested lesions total score ≤ 2 points; Active lesions total score > 2 points.
4th Caries activity assessment score | 6 months after baseline
  The activity of the clinically identified caries lesions (active/arrested) will be based on:
  Localisation of the lesion (No plaque stagnation area = 0, Plaque stagnation area = 1); Colour of the lesion (Brownish = 0; Whitish = 1); Feeling with probe (Lesion Smooth = 0; Lesion Rough = 1); No breakdown/breakdown on enamel surface: (No breakdown, or breakdown with smooth border area = 0; Breakdown with rough border area = 1); In case of gingival or proximal lesions (Healthy gingiva = 0; Bleeding on probing = 1).
  Arrested lesions total score ≤ 2 points; Active lesions total score > 2 points.
5th Caries activity assessment score | 8 months after baseline
  The activity of the clinically identified caries lesions (active/arrested) will be based on:
  Localisation of the lesion (No plaque stagnation area = 0, Plaque stagnation area = 1); Colour of the lesion (Brownish = 0; Whitish = 1); Feeling with probe (Lesion Smooth = 0; Lesion Rough = 1); No breakdown/breakdown on enamel surface: (No breakdown, or breakdown with smooth border area = 0; Breakdown with rough border area = 1); In case of gingival or proximal lesions (Healthy gingiva = 0; Bleeding on probing = 1).
  Arrested lesions total score ≤ 2 points; Active lesions total score > 2 points.
1st Clinical plaque score | Baseline
  Clinical plaque index ad modem Løe & Silness (1963) on selected teeth: 6+, 3+, 1+, +2, +4, +7, 7-,5-, 2-, -1, -3, -6.
  Clinical plaque score: 0 (No plaque visible), 1 (A film of plaque visible when using the probe), 2 (Moderate plaque accumulation that can be seen with the naked eye), 3 (An extensive plaque accumulation).
2nd Clinical plaque score | 1.5 months after baseline
  Clinical plaque index ad modem Løe & Silness (1963) on selected teeth: 6+, 3+, 1+, +2, +4, +7, 7-,5-, 2-, -1, -3, -6.
  Clinical plaque score: 0 (No plaque visible), 1 (A film of plaque visible when using the probe), 2 (Moderate plaque accumulation that can be seen with the naked eye), 3 (An extensive plaque accumulation).
3rd Clinical plaque score | 3 months after baseline
  Clinical plaque index ad modem Løe & Silness (1963) on selected teeth: 6+, 3+, 1+, +2, +4, +7, 7-,5-, 2-, -1, -3, -6.
  Clinical plaque score: 0 (No plaque visible), 1 (A film of plaque visible when using the probe), 2 (Moderate plaque accumulation that can be seen with the naked eye), 3 (An extensive plaque accumulation).
4th Clinical plaque score | 6 months after baseline
  Clinical plaque index ad modem Løe & Silness (1963) on selected teeth: 6+, 3+, 1+, +2, +4, +7, 7-,5-, 2-, -1, -3, -6.
  Clinical plaque score: 0 (No plaque visible), 1 (A film of plaque visible when using the probe), 2 (Moderate plaque accumulation that can be seen with the naked eye), 3 (An extensive plaque accumulation).
5th Clinical plaque score | 8 months after baseline
  Clinical plaque index ad modem Løe & Silness (1963) on selected teeth: 6+, 3+, 1+, +2, +4, +7, 7-,5-, 2-, -1, -3, -6.
  Clinical plaque score: 0 (No plaque visible), 1 (A film of plaque visible when using the probe), 2 (Moderate plaque accumulation that can be seen with the naked eye), 3 (An extensive plaque accumulation).
1st Clinical gingiva score | Baseline
  Clinical gingival index ad modem Løe & Silness (1963) on selected teeth: 6+, 3+, 1+, +2, +4, +7, 7-,5-, 2-, -1, -3, -6.
  Clinical gingiva score: 0 (Sound gingiva), 1 (A slight redness of the gingiva, no bleeding when probed), 2 (Bleeding when probed), 3 (Spontaneous bleeding).
2nd Clinical gingiva score | 1.5 months after baseline
  Clinical gingival index ad modem Løe & Silness (1963) on selected teeth: 6+, 3+, 1+, +2, +4, +7, 7-,5-, 2-, -1, -3, -6.
  Clinical gingiva score: 0 (Sound gingiva), 1 (A slight redness of the gingiva, no bleeding when probed), 2 (Bleeding when probed), 3 (Spontaneous bleeding).
3rd Clinical gingiva score | 3 months after baseline
  Clinical gingival index ad modem Løe & Silness (1963) on selected teeth: 6+, 3+, 1+, +2, +4, +7, 7-,5-, 2-, -1, -3, -6.
  Clinical gingiva score: 0 (Sound gingiva), 1 (A slight redness of the gingiva, no bleeding when probed), 2 (Bleeding when probed), 3 (Spontaneous bleeding).
4th Clinical gingiva score | 6 months after baseline
  Clinical gingival index ad modem Løe & Silness (1963) on selected teeth: 6+, 3+, 1+, +2, +4, +7, 7-,5-, 2-, -1, -3, -6.
  Clinical gingiva score: 0 (Sound gingiva), 1 (A slight redness of the gingiva, no bleeding when probed), 2 (Bleeding when probed), 3 (Spontaneous bleeding).
5th Clinical gingiva score | 8 months after baseline
  Clinical gingival index ad modem Løe & Silness (1963) on selected teeth: 6+, 3+, 1+, +2, +4, +7, 7-,5-, 2-, -1, -3, -6.
  Clinical gingiva score: 0 (Sound gingiva), 1 (A slight redness of the gingiva, no bleeding when probed), 2 (Bleeding when probed), 3 (Spontaneous bleeding).

CONTACTS AND LOCATIONS:
Overall Officials: Kim R. Ekstrand, ph.d, Study Chair — Institute of Odontology, University of Copenhagen
Locations (1):
- Institute of Odontology, University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Michou S, Benetti AR, Vannahme C, Hermannsson PG, Bakhshandeh A, Ekstrand KR. Development of a Fluorescence-Based Caries Scoring System for an Intraoral Scanner: An in vitro Study. Caries Res. 2020;54(4):324-335. doi: 10.1159/000509925. Epub 2020 Oct 14. PMID 33053552
- [Background] Kassebaum NJ, Bernabe E, Dahiya M, Bhandari B, Murray CJ, Marcenes W. Global burden of untreated caries: a systematic review and metaregression. J Dent Res. 2015 May;94(5):650-8. doi: 10.1177/0022034515573272. Epub 2015 Mar 4. PMID 25740856
- [Background] Pitts NB, Zero DT, Marsh PD, Ekstrand K, Weintraub JA, Ramos-Gomez F, Tagami J, Twetman S, Tsakos G, Ismail A. Dental caries. Nat Rev Dis Primers. 2017 May 25;3:17030. doi: 10.1038/nrdp.2017.30. PMID 28540937
- [Background] Bellini HT, Arneberg P, von der Fehr FR. Oral hygiene and caries. A review. Acta Odontol Scand. 1981;39(5):257-65. doi: 10.3109/00016358109162287. PMID 7039213
- [Background] Lussi A, Hibst R, Paulus R. DIAGNOdent: an optical method for caries detection. J Dent Res. 2004;83 Spec No C:C80-3. doi: 10.1177/154405910408301s16. PMID 15286128
- [Background] de Josselin de Jong E, Sundstrom F, Westerling H, Tranaeus S, ten Bosch JJ, Angmar-Mansson B. A new method for in vivo quantification of changes in initial enamel caries with laser fluorescence. Caries Res. 1995;29(1):2-7. doi: 10.1159/000262032. PMID 7867045
- [Background] LOE H, SILNESS J. PERIODONTAL DISEASE IN PREGNANCY. I. PREVALENCE AND SEVERITY. Acta Odontol Scand. 1963 Dec;21:533-51. doi: 10.3109/00016356309011240. No abstract available. PMID 14121956
- See also: Intraoral scanner featuring transillumination for proximal caries detection. An in vitro validation study on permanent posterior teeth — https://doi.org/10.1016/j.jdent.2021.103841